CLINICAL TRIAL: NCT01316094
Title: Long-term Study of ASP1941 - Long-term Study in Patients With Type 2 Diabetes Mellitus With Decreased Renal Function (Japanese)
Brief Title: A Study to Assess Efficacy and Safety of ASP1941 in Diabetic Patients With Renal Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1941-CL-0072
Record Dates: First submitted 2011-03-14; First posted 2011-03-16 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Pharmacokinetics; ASP1941; Renal impairment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency | interventions — ipragliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP group (Experimental): oral
  Interventions: Drug: ASP1941
- placebo group (Placebo Comparator): oral
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ASP1941 — oral
  Arms: ASP group
Drug: placebo — oral
  Arms: placebo group

SUMMARY:
This study is to assess the effect of renal function on the efficacy and safety of ASP1941 in type 2 diabetic patients with mild to moderate renal impairment.

DETAILED DESCRIPTION:
This study will be conducted in patients with type 2 diabetes mellitus and mild to moderate renal impairment who have inadequate glycemic control on an exercise program and stable diet, or one oral hypoglycemic agent.

The severity of the reduction in renal function in each subject will be classified according to the glomerular filtration rate (GFR) estimated using the Japanese GFR estimation equation. Subjects will start with a screening period, followed by a single-blind placebo run-in period, and will be randomized to the ASP1941 groups or the placebo group at a ratio of 2:1. For randomization, subjects will be stratified according to the severity of the reduction in renal function. In a treatment period, subject will receive study drug or placebo for 24 weeks under double-blind conditions.

At 24 week, subjects who are willing to continue participation in the study will receive study drug for another 28 weeks in an open label condition. ASP1941 can be increased. After completion of the study drug administration, a follow-up period will be provided.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus patient
* subject has been on an exercise program and stable diet, or one oral hypoglycemic agent (alpha-glucosidase inhibitor, sulfonylurea agent and pioglitazone)
* estimated GFR value based on the Japanese GFR estimation equation of ≥ 30 mL/min/1.73 m2 and < 90 mL/min/1.73 m2
* HbA1C value between 6.5 and 8.5%
* body mass index (BMI) 29.0 - 45.0 kg/m2

Exclusion Criteria:

* type 1 diabetes mellitus patients
* proliferative diabetic retinopathy
* subject has received insulin within 12 weeks before the study
* subject has a chronic disease which requires the continuous use of adrenocortical steroids, immunosuppressant, and loop diuretic
* serum creatinine > upper limit of normal
* proteinuria (albumin/creatinine ratio > 300mg/g)
* dysuria and/or urinary tract infection, genital infection
* significant renal, hepatic or cardiovascular diseases
* severe gastrointestinal diseases

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2011-01-18 (Actual); Primary Completion 2012-11-28 (Actual); Study Completion 2012-11-28 (Actual)

PRIMARY OUTCOMES:
changes in Hemoglobin A1c (HbA1c) | baseline and 24 weeks

SECONDARY OUTCOMES:
changes in fasting plasma glucose | baseline and 24 weeks
changes in fasting serum insulin level | baseline and 24 weeks
changes in eGFR (estimated glomerular filtration rate) | baseline and 52 weeks
safety assessed by the incidence of adverse events, vital signs, laboratory tests and 12-lead ECGs | for 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Shikoku
  - Tōhoku

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Kashiwagi A, Shestakova MV, Ito Y, Noguchi M, Wilpshaar W, Yoshida S, Wilding JPH. Safety of Ipragliflozin in Patients with Type 2 Diabetes Mellitus: Pooled Analysis of Phase II/III/IV Clinical Trials. Diabetes Ther. 2019 Dec;10(6):2201-2217. doi: 10.1007/s13300-019-00699-8. Epub 2019 Oct 12. PMID 31606880
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=91